CLINICAL TRIAL: NCT07199647
Title: Pain Beliefs, Spiritual Well-Being, and Health Beliefs on Complementary and Alternative Medicine in Rehabilitation Outpatients: A Cross-Sectional Study
Brief Title: Pain and Health Beliefs in Rehabilitation Outpatients
Status: Completed | Type: Observational
Sponsor: Gulseren Demir Karakilic (Other)
Responsible Party: Sponsor-Investigator, Gulseren Demir Karakilic, Assistant Professor, Principal Investigator, Bozok University
Organization: Bozok University (Other)
Other Study IDs: 2024-GOKAEK-2415_2024.12.18_29
Record Dates: First submitted 2025-09-22; First posted 2025-09-30 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Chronic Pain; Musculoskeletal Diseases
Keywords: Pain Beliefs; Spiritual Well-Being; Complementary and Alternative Medicine; Health Beliefs; Rehabilitation; Physical Medicine and Rehabilitation; Outpatients; Anxiety; Depression; Rehabilitation outpatients
MeSH Terms: conditions — Chronic Pain; Musculoskeletal Diseases; Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Rehabilitation Outpatients: Adult patients (18-65 years) attending a university hospital Physical Medicine and Rehabilitation outpatient clinic. Participants were evaluated once using self-report questionnaires and scales
  Interventions: Other: Questionnaire Administration

INTERVENTIONS:
Other: Questionnaire Administration — Participants completed a sociodemographic questionnaire, the Hospital Anxiety and Depression Scale, the Pain Beliefs Questionnaire, the Complementary, Alternative, and Conventional Medicine Attitude Scale, the Complementary and Alternative Medicine Health Belief Scale, and the Three-Factor Spiritual Well-Being Scale.

SUMMARY:
This cross-sectional study was conducted to investigate the relationships between patients' pain beliefs, health beliefs about complementary and alternative medicine, and levels of spiritual well-being in a Physical Medicine and Rehabilitation outpatient clinic. Adult participants between 18 and 65 years of age were enrolled. Standardized questionnaires were used to evaluate psychological status, pain-related beliefs, attitudes toward complementary and alternative medicine, and spiritual well-being. The study aimed to contribute to holistic pain management approaches by integrating psychological, spiritual, and health belief perspectives.

DETAILED DESCRIPTION:
Detailed Description:

This cross-sectional analytical study was designed to evaluate the interrelationships between pain beliefs, health beliefs regarding complementary and alternative medicine (CAM), and spiritual well-being in patients attending a Physical Medicine and Rehabilitation (PMR) outpatient clinic.

Rationale:

Chronic musculoskeletal pain is among the most frequent reasons for PMR admission. Prior research has examined pain beliefs, CAM utilization, or spirituality separately, yet little is known about their combined influence on patient coping, psychological status, and treatment orientation. Understanding these multidimensional factors is essential for advancing holistic, patient-centered rehabilitation strategies.

Study Design and Methods:

The study was conducted at Yozgat Bozok University, Faculty of Medicine, Department of PMR. A cross-sectional analytical design was employed. Eligible participants were adults aged 18-65 years who were literate, cognitively intact, and consented voluntarily. Exclusion criteria included communication or cognitive impairments, refusal to participate, or age outside the inclusion range.

Assessments:

Participants completed standardized, validated Turkish versions of the following instruments:

Hospital Anxiety and Depression Scale (HADS): evaluation of anxiety and depression symptoms.

Pain Beliefs Questionnaire (PBQ): assessment of organic and psychological pain beliefs.

Complementary, Alternative, and Conventional Medicine Attitude Scale (CACMAS): evaluation of attitudes toward CAM and conventional medicine.

Complementary and Alternative Medicine Health Belief Questionnaire (CHBQ): assessment of CAM-related health beliefs.

Three-Factor Spiritual Well-Being Scale (TFSWBS): measurement of transcendence, harmony with nature, and anomie.

Statistical Plan:

Descriptive statistics were calculated for demographic and clinical variables. Group comparisons were performed using Student's t-test, ANOVA, or chi-square tests, as appropriate. Correlation analyses explored associations among psychological, cognitive, and spiritual outcomes. Multiple regression models were applied to identify predictors of CAM health beliefs and spiritual well-being. Sample size was determined a priori using G*Power (version 3.1.9.7) to achieve 95% power with five predictors at α = 0.05.

Expected Contribution:

By integrating cognitive, psychological, and spiritual dimensions, the study seeks to clarify how pain beliefs and CAM health beliefs relate to spiritual well-being in rehabilitation patients. Findings are expected to support the incorporation of structured spiritual assessments and evidence-based CAM counseling into PMR practice to enhance holistic pain management.

ELIGIBILITY:
Inclusion Criteria:

* Adults between 18 and 65 years of age
* Attending the Physical Medicine and Rehabilitation outpatient clinic
* Able to read and write
* Cognitively intact
* Voluntarily willing to participate and able to provide informed consent

Exclusion Criteria:

* Younger than 18 years or older than 65 years
* Illiterate individuals
* Individuals with cognitive impairment
* Individuals with communication difficulties
* Patients who declined to participate or had incomplete data

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients aged 18 to 65 years who attended the Physical Medicine and Rehabilitation outpatient clinic of a university hospital in Türkiye.
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2024-12-19 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Pain Beliefs Questionnaire | At enrollment
  Description: The Pain Beliefs Questionnaire was developed in 1992 by Edwards and colleagues. It contains 12 items. Six items assess organic pain beliefs (score range: 6-30) and four items assess psychological pain beliefs (score range: 4-20). Participants rate each item using a Likert-type scale from 1 to 5. Higher scores on the organic subscale indicate stronger beliefs in an organic cause of pain (considered maladaptive), while higher scores on the psychological subscale indicate stronger beliefs in a psychological origin of pain (considered more adaptive).
Three-Factor Spiritual Well-Being Scale | At enrollment
  Description: The Three-Factor Spiritual Well-Being Scale was developed in 2017 by Eksi and Kardas. It contains 29 items with three subscales: transcendence (11 items, score range: 11-55), harmony with nature (6 items, score range: 6-30), and anomie (12 items, score range: 12-60; reverse-scored). Items are rated on a 5-point Likert scale. The total score ranges from 29 to 145. Higher total scores indicate greater levels of spiritual well-being (a better outcome).
Complementary and Alternative Medicine Health Belief Scale | At enrollment
  This scale was developed in 2004 by Lie and Boker. It contains 10 items. Each item is scored on a seven-point Likert scale. Three of the items are reverse-scored. The total score ranges from 10 to 70. Higher scores indicate stronger health beliefs related to complementary and alternative medicine. The scale does not have a cut-off score.

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale | At enrollment
  This scale was developed in 1983 by Zigmond and Snaith. It contains 14 items. Seven items measure anxiety and seven items measure depression. Each item is scored on a scale from 0 to 3. Some items are reverse-scored. The cut-off score is 10 for anxiety and 7 for depression. Higher scores indicate higher levels of anxiety or depression. The scale does not provide a total score but gives separate scores for the two subscales.
Complementary, Alternative, and Conventional Medicine Attitude Scale | At enrollment
  This scale was developed in 2010 by McFadden and colleagues. It contains 25 items. It has three subscales: attitudes toward complementary and alternative medicine, dissatisfaction with conventional medicine, and holistic balance. Participants rate each item using a Likert-type scale. The scale does not have a cut-off score. Higher scores indicate a more favorable attitude toward complementary and alternative medicine and stronger belief in holistic balance.

CONTACTS AND LOCATIONS:
Overall Officials: Gülseren Demir Karakılıç, Asst Prof, Principal Investigator — Yozgat Bozok University
Locations (1):
- Yozgat Bozok University Faculty of Medicine, Department of Physical Medicine and Rehabilitation, Yozgat, Yozgat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated and analyzed during the current study are available from the corresponding author on reasonable request. De-identified data will be shared for academic and research purposes in accordance with institutional and ethical guidelines.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: De-identified individual participant data and supporting documents will be available beginning 6 months after publication of the study results and will remain available for 5 years.
Access Criteria: De-identified individual participant data and supporting documents will be available upon reasonable request to the corresponding author for academic and research purposes only. Requests will be reviewed by the study investigators, and data will be shared via secure electronic transfer in accordance with institutional and ethical guidelines.
URL: https://bozok.edu.tr

REFERENCES:
- [Background] Uslu, F. (2020). Geleneksel ve tamamlayıcı tıp (getat) sağlık inanış anketinin türkçe geçerlilik ve güvenilirlik çalışması. (Uzmanlık Tezi). Sağlık Bilimleri Üniversitesi Ankara Dışkapı Yıldırım Beyazıt Sağlık Uygulama ve Araştırma Merkezi Aile Hekimliği Kliniği, Ankara. https://tez.yok.gov.tr/UlusalTezMerkezi/ sayfasından erişilmiştir. (Tez Numarası 644233).
- [Background] Elif, K. Ö. S. E., Hasan Çetin Ekerbiçer, and Ünal Erkorkmaz. "Complementary, alternative and conventional medicine attitude scale: Turkish validity reliability study." Sakarya Tıp Dergisi 8.4 (2018): 726-736.
- [Background] Hyland ME, Lewith GT, Westoby C. Developing a measure of attitudes: the holistic complementary and alternative medicine questionnaire. Complement Ther Med. 2003 Mar;11(1):33-8. doi: 10.1016/s0965-2299(02)00113-9. PMID 12667973
- [Background] Edwards LC, Pearce SA, Turner-Stokes L, Jones A. The Pain Beliefs Questionnaire: an investigation of beliefs in the causes and consequences of pain. Pain. 1992 Dec;51(3):267-272. doi: 10.1016/0304-3959(92)90209-T. PMID 1491853
- [Background] Aydemir, O. J. T. P. D: Hastane Anksiyete ve Depresyon Ölçeği Türkçe Formunun Geçerlilik ve Güvenilirliği. Türk Psikiyatri Dergisi, 8, 187-280, 1997.
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Okan N, Kose N, Kardas S. Spiritual Contradiction Scale: A New Way of Understanding Internal and External Contradictions. J Relig Health. 2024 Apr;63(2):1567-1584. doi: 10.1007/s10943-023-01924-2. Epub 2023 Oct 11. PMID 37819529
- [Background] Berk HO, Bahadir G. [The experience of chronic pain and pain beliefs]. Agri. 2007 Oct;19(4):5-15. Turkish. PMID 18159574